CLINICAL TRIAL: NCT02497664
Title: Optimizing (Breathing) Techniques for Radiotherapy of Esophageal and Lung Carcinomas
Acronym: ABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RT2015-04
Record Dates: First submitted 2015-06-22; First posted 2015-07-14 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Esophageal Cancer; Lung Cancer
Keywords: Radiotherapy; Active Breathing Control Technique
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active Breathing Control (Other): Planning-CT will be made of patients using the Active Breathing Control Technique (in expiration and inspiration phase)
  Interventions: Other: Active Breathing Control

INTERVENTIONS:
Other: Active Breathing Control

SUMMARY:
Neo-adjuvant chemoradiotherapy (neo-CRT) is increasingly applied in the curative treatment of esophageal cancer, with the aim to downstage the tumor, to increase the rate of radical resections, and consequently to improve the survival rates. Due to improved survival, it will become increasingly important to minimize the radiation-induced toxicity among long-term survivors.

In the management of locally advanced non small cell lung cancer (NSCLC), radiotherapy is the standard treatment modality. However, the dose that can be safely applied to the tumour is limited by the risk of cardiac and pulmonary complications, which even led to decreased survival in a randomised study, when a higher tumor dose was administered [1].

Radiation induced pulmonary and cardiac toxicity are the most important late side effects after thoracic radiotherapy [2-4].

The aim of this study is to reduce the radiation dose of heart (and lungs) in order to reduce the toxicity risk.

In recent years, the active breathing control (ABC) technique has been introduced in the radiotherapy for left sided breast cancer patients, to minimize the radiation dose to the heart. These patients are irradiated in the inspiration phase, in which the distance between the heart and the breast is largest, while the lungs extend.

Breath hold might also be beneficial for radiotherapy of esophageal and lung tumors. For these patients the expiratory phase might theoretically be more beneficial to reduce the heart dose. However, the inspiration phase might be better for the dose to the lungs, which consequently allows cardiac dose reduction.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven esophageal cancer (adeno-, or squamous cell carcinoma) of the mid or distal esophagus or stage III NSCLC (any histological subtype).
* Scheduled for external-beam photon radiotherapy with curative intention.
* WHO 0-2.
* Age >= 18 years
* Written informed consent.

Exclusion Criteria:

* Serious respiratory distress
* Noncompliance with any of the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Mean Hart Dose (MHD) | At 6 weeks after start of radiation therapy

SECONDARY OUTCOMES:
Mean Lung Dosis (MLD) | At 6 weeks after start of radiation therapy
Position of the heart in relation to the target volumes | At 6 weeks after start of radiation therapy
Internal Target Volume (ITV) margin (margin for breathing movement defined as ITV - Gross Tumor Volume (GTV)) | At 6 weeks after start of radiation therapy
Dose Volume Histogram (DVH) parameters of the heart | At 6 weeks after start of radiation therapy
  V5, V10, V20, V30, V40, V50, V60

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands